CLINICAL TRIAL: NCT07307755
Title: Application of the Validity and Reliability of the Modified O'Sullivan Functional Balance (mOFB) Test in Multiple Sclerosis Patients
Brief Title: The Validity and Reliability of the Modified O'Sullivan Functional Balance (mOFB) Test for Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, Sanko University, Sanko University
Other Study IDs: hakanpolat8
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: MULTİPLE SCLEROSİS; BALANCE; VALİDİTY; RELİABİLİTY
Keywords: MULTİPLE SCLEROSİS; BALANCE; VALİDİTY; RELİABİLİTY
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the validity and reliability of the Modified O'Sullivan Functional Balance (OFB) Test, which is used to assess balance in individuals diagnosed with Multiple Sclerosis (MS).

Multiple Sclerosis is a chronic nervous system disease that can cause symptoms such as balance problems, difficulty walking, and fatigue, which negatively affect daily life. Balance disorders are common in MS patients, increasing the risk of falls and leading to a decrease in physical activity levels. Therefore, the accurate and reliable assessment of balance in MS patients is of great importance.

This study will include volunteer MS patients treated at the Physical Therapy and Rehabilitation Department of SANKO University Sani Konukoğlu Application and Research Hospital who meet the inclusion criteria. After recording the participants' demographic and disease-related information, their balance, body control, and walking skills will be assessed using various clinical tests. These tests include the Berg Balance Test, Mini-BESTest, O'Sullivan Functional Balance Test, Modified O'Sullivan Functional Balance Test, Trunk Instability Scale, and L Test.

Assessments will be conducted taking into account the fatigue commonly seen in MS patients, and participants will be allowed to rest when needed. The results obtained will reveal whether the Modified O'Sullivan Functional Balance Test is a reliable and applicable method for assessing balance in MS patients.

It is anticipated that the results of this study will contribute to clinical practice in the assessment of balance in MS patients and assist in the more effective planning of the rehabilitation process.

DETAILED DESCRIPTION:
This study is a methodological research designed to evaluate the validity and reliability of the Modified O'Sullivan Functional Balance (OFB) Test in individuals diagnosed with Multiple Sclerosis (MS).

Before the assessments, all participants will receive a practical explanation and demonstration of how each test is performed. Considering the high prevalence of fatigue in individuals with MS, the assessment protocol will be planned to allow adequate rest periods, and participants will be seated and rested prior to the administration of the Modified O'Sullivan Functional Balance (OFB) Test.

Assessments will be conducted on two separate days with a one-week interval, consisting of two sessions per day. On the first day, during the first session, the Modified O'Sullivan Functional Balance (OFB) Test will be administered by the first assessor (Dr. PT Meltem Uzun). In the same session, the Berg Balance Scale, Mini-BESTest, Trunk Impairment Scale, and L Test will also be applied. During the second session on the first day, the Modified O'Sullivan Functional Balance (OFB) Test will be administered by the second assessor (Dr. PT Hakan Polat).

On the second assessment day, the Modified O'Sullivan Functional Balance (OFB) Test will be administered sequentially by Dr. PT Meltem Uzun and Dr. PT Hakan Polat. This assessment protocol will allow the evaluation of both inter-rater reliability and test-retest reliability by performing the same measurements on different days and by different physiotherapists.

All assessments will be carried out in the Application and Research Laboratory of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, SANKO University. Participants will be evaluated in the same environment during all sessions to minimize the effects of environmental factors on performance. The assessment room will be maintained at normal room temperature, adequately illuminated, and have a firm surface floor. Each assessment session will last approximately 25-30 minutes, while the total duration of the first session, including interviews and evaluations, will be approximately 40-45 minutes.

Prof. Dr. Suat Erel and Assoc. Prof. Dr. Emel Taşvuran Horata will be responsible for the planning of the study, formulation of hypotheses, interpretation of results, and preparation of the scientific manuscript.

All collected data will be coded using project identification numbers to ensure participant confidentiality. Data will be stored and managed using Microsoft Excel, and access will be restricted exclusively to the research team members involved in the project.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-65 years
* Volunteers participating in the study
* Individuals not using any assistive devices
* Individuals unable to maintain the tandem stance test for more than 10 seconds
* Individuals with an Expanded Disability Status Scale (EDSS) score ≤ 5.5

Exclusion Criteria:

* Pregnant or within the first 3 months postpartum
* Received corticosteroid treatment within the last month
* Took any medication affecting walking ability within the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Neurology Outpatient Clinic of SANKO University Sani Konukoğlu Application and Research Hospital with a diagnosis of Multiple Sclerosis
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-14 (Actual)

PRIMARY OUTCOMES:
Modified O'Sullivan Functional Balance (mOFB) Test | 1 YEARS
  The mOFB is a modified version of the OFB that incorporates adjusted grading criteria, combined with external resistance to challenge static balance and weight shifting to challenge dynamic balance. A previous study found that this modified test had low to moderate reliability due to the lack of clear test instructions and scoring criteria. To address these limitations, we developed standardised test instructions and scoring criteria, as summarised in the Supplementary Material , before evaluating the psychometric properties of the mOFB. The assessment takes approximately 5 minutes and can be performed on a fixed bed or chair using only a stopwatch. The test condition consists of static sitting balance, dynamic sitting balance, static standing balance, and dynamic standing balance. Scoring is based on observing the patient's ability to maintain balance while sitting or standing quietly for 60 seconds, respond to external disturbances, and reach in various directions beyond
O'Sullivan Functional Balance Test | 1 YEARS
  The OFB is a scoring tool used to assess both static and dynamic balance in various positions. This test highlights the ability to maintain postural stability and make postural adjustments in response to voluntary movements such as turning the head or torso, reaching for an object on the ground, and shifting body weight. The OFB test uses a 5-level ordinal rating scale: zero, poor, fair, good, and normal. A zero score indicates an inability to maintain balance, while a 'normal' score reflects normal balance performance . This study converted the rating scale into sequential scores ranging from 0 to 4, where 0 indicates an inability to maintain balance independently and 4 indicates normal balance, assessed across four components: static sitting balance, dynamic sitting balance, static standing balance, and dynamic standing balance. The total OFB score is 16, and sub-scores can be given for individual test positions. For example, the static sitting balance sub-score ranges from 0 to 4.
Berg Balance Scale (BBS) | 1 YEARS
  The BBS is widely used and is currently accepted as the reference standard for assessing balance in individuals who have suffered a stroke. The BBS consists of 14 functional balance tasks that focus on the ability to maintain a position and make postural adjustments based on voluntary movements. It is simple to administer and requires minimal equipment and time to complete. Each item is scored between 0 and 4; 0 indicates inability to perform the task, while 4 indicates optimal performance. The maximum score is 56, and scores below 45 indicate a high risk of falling.
Trunk Impairment Scale (TIS) | 1 YEARS
  The Trunk Impairment Scale (TIS) is designed to measure motor impairment of the trunk by assessing static and dynamic sitting balance and trunk coordination. The original TIS assesses three components: static sitting balance (maximum score = 7), dynamic sitting balance (maximum score = 10), and trunk coordination (maximum score = 6), with a total of 23 points possible. A key advantage of the TIS is its minimal equipment requirement, making it highly practical for use in clinical settings.
L test | 1 YEARS
  This test indirectly assesses walking speed and dynamic balance during walking and turning activities. It is a modified version of the TUG test. The walking path is L-shaped. The L test is a more comprehensive test than the TUG test as it involves a greater walking distance and turning activity in both directions. The L test assesses the fundamental components of functional mobility, such as balance, transfer, walking, and turning. During the test, the individual stands up from the chair, walks 3 metres, turns right, walks 7 metres, then turns back and walks along the same path to sit down on the chair. The measured distance will be recorded in metres.
Mini Best Test | 1 YEARS
  This is one of the clinical tests used to assess walking and balance. It consists of four sub-parameters: preparatory movement, reactive postural control, sensory orientation, and dynamic walking, comprising a total of 14 items. It is a test scored out of a total of 28 points, taking an average of 10-15 minutes to complete. A high score indicates high function.

CONTACTS AND LOCATIONS:
Overall Officials: HAKAN POLAT, phd, Study Director — Sanko University
Locations (1):
- Sanko Unıversıty, Gaziantep, şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
will be decided when the study is completed